CLINICAL TRIAL: NCT03759886
Title: Mechanical Bowel Preparation and Oral Antibiotic Prophylaxis vs. Mechanical Bowel Preparation in Colorectal Surgery With i.v. Antibiotic Prophylaxis
Brief Title: Oral Antibiotic Prophylaxis in Colorectal Surgery
Acronym: ABCR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Dr. Boris Jansen-Winkeln, Consultant Colorectal Surgery, University of Leipzig
Other Study IDs: ABCR
Record Dates: First submitted 2018-10-16; First posted 2018-11-30 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Surgical Site Infection; Anastomotic Leak
MeSH Terms: conditions — Surgical Wound Infection; Anastomotic Leak | interventions — Metronidazole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral Antibiotics: The patients get mechanical bowel preparation and oral antibiotic prophylaxis with 4g Paromomycin (Paromomycin Sulfate Powder) and 1 g Metronidazole p.o. and perioperative i.v. antibiotic prophylaxis with Ertepanem 1g i.v.
  Interventions: Drug: Paromomycin Sulfate Powder
- iv Antibiotics: The patients get mechanical bowel preparation and perioperative i.v. antibiotic prophylaxis with Ertepanem 1g i.v.

INTERVENTIONS:
Drug: Paromomycin Sulfate Powder — The patients receive Paromomycin and Metronidazole the day prior to colorectal surgery after mechanical bowel preparation
  Other Names: Metronidazole
  Groups: Oral Antibiotics

SUMMARY:
The investigators perform a case-control study to compare preparation before elective colorectal surgery. The first group is a prospective patient - registry in all patients with mechanical bowel preparation (MBP) and oral antibiotic prophylaxis the day before colorectal surgery. The second group is a historic collective of patients with MBP only and colorectal surgery. The cases were matches in American Society of Anesthesiologists (ASA) physical status classification system, BMI, operative procedure and risk factors.

ELIGIBILITY:
Inclusion Criteria:

* all colorectal resections

Exclusion Criteria:

* allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients wich receive elective colorectal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infections | 30 days (exact 30 days after the Operation date)
  Any kind of surgical site infection in the postoperative course.

SECONDARY OUTCOMES:
Anastomotic Leak | 30 days (exact 30 days after the Operation date)
  All with objective methods proven anastomotic leakage (like contrast enema, re-operation or endoscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Jansen-Winkeln, PD Dr., Principal Investigator — University of Leipzig
Locations (1):
- Universitätsklinikum Leipzig - AöR, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mehdorn M, Lubbert C, Chaberny IF, Gockel I, Jansen-Winkeln B. Mechanical plus oral bowel preparation with paromomycin and metronidazole reduces infectious complications in elective colorectal surgery: a matched case-control study. Int J Colorectal Dis. 2021 Sep;36(9):1839-1849. doi: 10.1007/s00384-021-03931-9. Epub 2021 Apr 25. PMID 33895874